CLINICAL TRIAL: NCT07337343
Title: Co-Development and Validation of Colonic Symptom Pictograms for Young People
Status: Not yet recruiting | Type: Observational
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Gayl Humphrey, Dr, University of Auckland, New Zealand
Other Study IDs: Colonic_Pictogram_Val
Record Dates: First submitted 2025-12-14; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Constipation - Functional; Abdominal Pain (AP); Nausea and Vomitting; Bloating; Flatulence; IBS, Constipation Predominant
Keywords: children and adolescents; pictograms; co-design; validation
MeSH Terms: conditions — Abdominal Pain; Nausea; Flatulence; Ichthyosis Bullosa of Siemens

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children and young people aged 8-17 years: children and young people aged 8-17 years with lower GI symptoms
  Interventions: Other: Pictogram comprehension and validation

INTERVENTIONS:
Other: Pictogram comprehension and validation — This study aims to codesign and validate Colonic Symptom Pictograms for use with Young People to support them in distinguishing and reporting the symptoms they experience.

SUMMARY:
Severe constipation affects 10% of children, often leading to significant physical and emotional distress. While constipation is commonly associated with impaired bowel movements, it is fundamentally linked to abnormalities in colonic motility - the coordinated contractions that facilitate passage of stool through the colon and out of the body. Diagnosis of constipation is based upon the Rome IV criteria, which assess symptoms as reported or remembered over the previous 3 months.

However, reporting symptoms experienced can be challenging for children and young people for many reasons, such as the overlap of sensations, including fullness, bloating, and discomfort, and an inability to recall or precisely distinguish and describe what they are feeling.

This study intends to design, develop, and validate symptom pictograms for children aged 8-17 with colonic or lower gut symptoms.

DETAILED DESCRIPTION:
Severe refractory constipation affects 10% of children, often leading to significant physical and emotional distress. While constipation is commonly associated with impaired bowel movements, it is fundamentally linked to abnormalities in colonic motility - the coordinated contractions that facilitate passage of stool through the colon and out of the body. Diagnosis of constipation is based upon the Rome IV criteria, which assess symptoms as reported or remembered over the previous 3 months.

However, reporting symptoms experienced can be challenging for children and young people for many reasons, such as an overlap of sensations, such as fullness, bloating, and discomfort, and an inability to recall or precisely distinguish and describe what they are feeling. An earlier study approved by the New Zealand Health and Disability Ethics Committee (HDEC reference 2022 FULL 12705) designed, developed, and validated a set of upper gastric symptom pictograms to help children and young people record their symptoms during a test called body surface gastric mapping (BSGM). The use of these symptom pictograms has enabled improved correlation of gastric activity with symptoms to assist in the diagnostic process.

This study intends to build on this knowledge and apply it to design, develop, and validate symptom pictograms for children aged 8-17 with colonic or lower gut symptoms.

Objective To co-design, develop, and validate a set of pictograms representing lower gastrointestinal (GI) symptoms that are easily understood and useful for children and young people aged 8-17 years. The pictograms will support improved symptom communication, enhance clinical assessment, and be evaluated for comprehension, acceptability, and utility during investigations.

Study Design and Methodology:

A multi-phase, mixed-methods study incorporating participatory co-design, iterative prototyping, and validation testing with children and young people aged 8-17 years.

Study Population Children and young people aged between 8-17-years with and without lower gastrointestinal symptoms.

Participant Numbers Phase One: A review of current guidelines and symptom questionnaires to confirm core colonic symptoms relevant to refractory constipation, and a web-based search for images depicting these symptoms to identify common concepts. Final selection will be confirmed by the research team and clinical advisors.

Phase Two: Co-design. A minimum of 30 children and young people.

Phase Three: Pictogram Development and Refinement based on Phase I, and check the designs for clarity with a group of young people before the validation phase.

Phase Four: Validation: At least 80 children and young people with and without lower gastrointestinal symptoms such as constipation.

Inclusion Criteria For all phases, the main inclusion criteria for all children and young people participants are that they are,

* aged between 8-17 years,
* able and willing to complete the tasks, and
* communicate in English or be supported by a caregiver, whānau (family), or responsible adult to participate

Criteria for Evaluation Phase One: Thematic analysis of symptom concepts and visual ideas, and identification of the symptoms that will be designed and presented visually

Phase Two: Gather pictures of symptoms drawn by young people. Review of symptom concepts drawn by participants, reviewing differences and similarities by different ages, sex, and ethnicity (as appropriate), such as facial expressions, colours, and prompts used. Design new colonic symptom pictograms that reflect the outcome of Phases One and Two.

Phase Three: Confirm the clarity and qualitative feedback on preferred styles and features of the new pictograms.

Phase Four: Following ISO standard 9186, Comprehension Validity (translucency and transparency) and content validity index metrics, the pictograms will be evaluated for understanding and agreement and validated against existing tools.

Statistical Methods Phases Two and Three: A convenience sample will be adopted, so no power analyses have been calculated.

Phase Four: The proposed minimum of 80 participants is expected to be sufficient to test the guessability, translucency, and validity of six to ten pictograms and provide precision about the mean and variance for the consistency, reliability, and construct validity. (Boateng et al. 2018)

Analysis Phase One: A review of common themes, symptom concepts, and visual ideas will be used to identify the relevant symptoms that need to be co-designed.

Phase Two: A review of the common themes, images, and prompts to enable new pictograms to be designed and developed

Phase Three: A review of the responses for each symptom pictogram recognition and understanding.

Phase Four: Descriptive and comparative statistics will be utilised. Translucency will be assessed using a visual analogue scale, ranging from 0 (complete lack of correlation) to 5 (very high correlation agreement). Achieving an agreement of ≥3 is identified as an acceptable level of correlation between the pictogram and its meaning. Validity will be evaluated using the Content Validation Index (CVI) and Pearson's correlation coefficient equations, with internal reliability assessed using Cronbach's α. A CVI greater than 80% and a coefficient level above 0.65 are acceptable.

ELIGIBILITY:
Inclusion Criteria:

Children and Young people are aged between 8-17 years,

* have lower gut or constipation symptoms,
* can communicate in English or be supported to participate by a caregiver, whānau, or other responsible person. Phase Four will include international invitations to participants with lower gut or constipation symptoms. Healthy volunteers will not be recruited.

Exclusion Criteria:

* Children and Young people with developmental or cognitive disorder that precludes their ability to understand the study,
* Children and Young people who do not have access to a digital device with internet connectivity,
* unable to read English,
* parent does not consent

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: International cohort of young people aged 5-17 years
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Validation of each Pictogram | Analyses will be undertaken once the last participant (80th) has completed the online survey. This is anticipated to occure 6 months fro start of the study,
  We hypothesize that the new colonic pictogram-based symptom reporting will demonstrate equivalent or superior validity and reliability compared to traditional questionnaire-based methods for reporting constipation symptoms in young people. Specific analyses will be to evaluate the pictograms for comprehension, translucency, face validity, construct validity, and convergent and divergent validity.
  * Comprehension: responses will be measured using a scale from 1= correct , 4= correct and 5 = did not answer.
  * Translucency: Likert rating scale to report how well participants report the pictograms reflect the intended symptoms Convergent: Using Rome IV Section B responses will be compared to the correct pictogram to assess correlations Divergent: A lower relationship between pictogram comprehension and PedsQL Oral Health questionnaire will be assessed Concurrent: PedQL answers will assess the association between accruated identifying the pictograms and health outcomes

IPD SHARING:
Plan to Share IPD: No
During the study, data may be collected from participants who identify, for example, as Māori (indigenous population of New Zealand). Providing insights and information to research is a tāonga (treasure) and will be treated accordingly. The research team aims to ensure data sovereignty in light of, for example, the global directives on Indigenous rights and local treaties such as Te Tiriti o Waitangi in Aotearoa/New Zealand. We will not routinely make IPD data available. However, we will consider requests where the proposal meets international guidelines to ensure that datasets are analysed according to the data governance of the respective cultures, such as Tikanga Māori in New Zealand.